CLINICAL TRIAL: NCT03777605
Title: Absorption and Pharmacokinetics of Nitroglycerin as a Tablet or in the Form of Rapidly Degradable Capsule in Young Healthy
Brief Title: Absorption and Pharmacokinetics of Nitroglycerin to a New Formulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Ole Winther Rasmussen, Clinical professor, Kolding Sygehus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nitroglycerine1523 (NTG1523)
Record Dates: First submitted 2018-12-03; First posted 2018-12-17 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Nitroglycerin

STUDY DESIGN:
Intervention Model Description: A randomized, cross over design
Masking Description: All tablets are processed, marked and coded by a pharmacist,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "NTG1523", rapid absorbable capsule (Experimental): Nitroglycerine 0.4 milligram taken as ordinary tablets or "NTG1523" rapid absorbable capsule once in the morning, and subsequently blood samples and observations for 2 hours are performed
  Interventions: Drug: Nitroglycerin 0.4 MG

INTERVENTIONS:
Drug: Nitroglycerin 0.4 MG — The study evaluate absorption rate of nitroglycerine 0.4 milligrams as tablets or a quickly absorbable capsuel "NTG1523" determined by T-max and area under the response curve in the blood of NTG as well as from clinical effects.
  Data is entered on data sheet in anonymous form and processed. The results are presented in anonymous form by publication and lecture. Experts are given the supplement: "The applicant's rights in a biomedical research project
  Other Names: "NTG1523"

SUMMARY:
The study evaluate the absorption rate of different sublingual formulation of nitroglycerine (NTG) either in the form of available tablets or a new rapid absorbable gelation capsule formulation "NTG1523" by determining T-max and area under the response curve of nitoglycerine in blood concentration as well as from clinical effects after intake. Data is entered on data sheet in anonymous form and processed. The results are presented in anonymous form by publication and lecture. Experts are given the supplement: "The applicant's rights in a biomedical research project

DETAILED DESCRIPTION:
Ten healthy young volunteers are recruited,, and the experiments begin at 07:45 after an overneight fast. BMI and blod pressure are recorded and a catheter is inserted in an anticubical vein for blood samples.

At 08.00 a sublingual tablet (Takeda, nitroglycerin 0.4 milligrams) tablet or a "NTG1523" capsule with 0.4 milligrams of nitroglycerine is placed under the tongue in random order. Subsequently, blood samples are taken every minute for 10 minutes, then every 10 minutes the following two hours. In addition, blood pressure and puls rate are measured every second minute the first ten minutes, and then every 10 minutes.Side effects and time to the participants registrate any effect of the drugs are assessed in a prefabricated scheme.

The disadvantages associated with the experiment are sought monitored by adverse event registration which ends at the end of the trial. The trial day lasts 2 hours in which blood samples are taken as described above, and blood pressure and records are stored .

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteers
* Must be able to swallow tablets

Exclusion Criteria:

* Insulin dependent diabetes
* Thyroid disease
* any medial treatment

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-12-23 (Estimated); Primary Completion 2020-12-05 (Estimated); Study Completion 2020-12-23 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration of Nitroglycerine as a tablet or in the form of rapidly degradable capsule "NTG1523" in young healthy controls | From 2 weeks up til 5 weeks
  Peak Plasma Concentration (Cmax)(ng(ml) of nitroglycerine

SECONDARY OUTCOMES:
Blood pressure in response to Nitroglycerine | From 2 weeks up til 5 weeks
  Blood pressure (mmHg)
Puls rate in response to Nitroglycerine | From 2 weeks up til 5 weeks
  puls rate (beat/min)

CONTACTS AND LOCATIONS:
Overall Officials: ole W Rasmussen, M.D. Dr.Sci, Principal Investigator — Medical Dept.,Kolding Hospital, SLB, Denmark
Locations (1):
- Kolfding Sygehus, SLB, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakashima E, Rigod JF, Lin ET, Benet LZ. Pharmacokinetics of nitroglycerin and its dinitrate metabolites over a thirtyfold range of oral doses. Clin Pharmacol Ther. 1990 May;47(5):592-8. doi: 10.1038/clpt.1990.80. PMID 2111749
- [Result] McAllister A, Mosberg H, Settlage JA, Steiner JA. Plasma levels of nitroglycerin generated by three nitroglycerin patch preparations, Nitradisc, Transiderm-Nitro and Nitro-Dur and one ointment formulation, Nitrobid. Br J Clin Pharmacol. 1986 Apr;21(4):365-9. doi: 10.1111/j.1365-2125.1986.tb05208.x. PMID 3085698